CLINICAL TRIAL: NCT00005926
Title: A Phase II Trial of Gemcitabine, Herceptin, and Radiation for Regionally Confined Adenocarcinoma of the Pancreas
Brief Title: Gemcitabine, Herceptin and Radiation to Treat Cancer of the Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000161; 00-C-0161
Record Dates: First submitted 2000-06-28; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-06

CONDITIONS: Pancreatic Cancer; Pancreatic Neoplasm
Keywords: Cancer; Gemzar; Her-2/Neu; Pancreatic; Radiotherapy; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Gemcitabine; Trastuzumab; Radiotherapy

INTERVENTIONS:
Drug: Gemcitabine
Drug: Herceptin
Procedure: Radiation therapy

SUMMARY:
This study will examine the safety and effectiveness of the drugs Gemcitabine and Herceptin, given in conjunction with radiation therapy, for treating patients with cancer of the pancreas. Gemcitabine is standard therapy for advanced pancreatic cancer. It damages tumor cells and may enhance the effects of radiation therapy. Herceptin is a genetically engineered antibody that has prevented some tumors from growing in patients with breast cancer. Because breast and pancreatic cancer cells share an characteristic related to how Herceptin works (similar HER-2/neu receptor proteins), it is thought that this drug may also inhibit growth of tumors of the pancreas.

Patients with pancreatic cancer may be eligible for this study. Candidates will be screened with a physical examination, chest X-ray, blood tests, electrocardiogram, and computerized tomography (CT) scan of the chest, abdomen and pelvis. They will also have a minor surgical procedure called a laparoscopy to evaluate the extent of their cancer. This procedure, done under general anesthesia, requires an overnight hospital stay. A small incision (about 1 inch) is made in the abdomen and a thin, flexible tube with a light and special fibers at the end is inserted into the opening. This device, called a laparoscope, allows the surgeon to see inside the abdominal cavity to evaluate the tumor and also to remove a small piece of tumor tissue for examination.

Patients accepted into the study will be assigned to one of two treatment groups, according to whether or not their tumor can be removed with surgery. Patients will be asked to complete a Quality of Life Evaluation before treatment begins and again at each follow-up visit. This 15-minute questionnaire assesses patients' feelings, their ability to carry out usual activities, and the effects of therapy on their general health and well being.

Patients in both treatment groups will be given the same chemotherapy, on an outpatient basis unless special circumstances require hospitalization. Gemcitabine is infused over 30 to 60 minutes through an intravenous catheter (IV)-a thin plastic tube inserted into an arm vein. Herceptin is then given over 30 to 90 minutes through the same IV line. Radiation therapy to the abdomen will start the same day, after the drugs have been administered, and will continue for the next 4 days. This treatment cycle-chemotherapy plus 5 days of radiation therapy-will be repeated each week for 6 weeks.

Within 6 weeks after the last treatment, the patient's tumor will be evaluated with a blood test and CT scan of the chest, abdomen and pelvis to determine if it can be removed with surgery. If so, the procedure will be done under general anesthesia and will require a 7- to 10-day hospital stay. If the tumor cannot be removed with surgery, another biopsy will be taken to evaluate the tumor's response to the chemotherapy and radiation treatment.

All patients will receive additional chemotherapy beginning 6 weeks after surgery (for patients whose tumors were removed) or 6 weeks after radiation therapy (for patients whose tumors could not be removed). Gemcitabine and Herceptin will be given IV once a week for 3 weeks followed by a week of rest. This 4-week treatment cycle will be repeated up to six times.

After treatment ends, patients will be evaluated with CT scans or X-rays and blood tests every 3 to 4 months for the first 2 years and every 6 months thereafter to evaluate disease status.

DETAILED DESCRIPTION:
This is a phase II study of gemcitabine and Herceptin given weekly as a bolus infusion administered concurrently with radiotherapy in patients with regionally confined resectable or unresectable adenocarcinoma of the pancreas that overexpress HER2. Patients will be treated with external beam radiation in a standard manner over 6 weeks prior to surgical exploration. Gemcitabine and Herceptin will be administered on the first day of irradiation and weekly during the course of radiotherapy. Patients will be assessed for resectability after treatment and may undergo a pancreatic resection. Patients will then be treated with once weekly gemcitabine and herceptin for three weeks followed by 1 week of rest for up to 6 months. Patients will be assessed clinically for toxicity, tumor response, progression-free survival, and overall survival.

ELIGIBILITY:
Patients must have regionally confined histologically or cytologically proven adenocarcinoma of the pancreas or Ampulla of Vater. Tumors must overexpress HER2 as demonstrated by greater than or equal to 2+ immunohistochemical staining of the biopsy specimen.

Patients must sign an informed consent.

Patients must have an ECOG performance status of less than or equal to 2.

Patients should have a serum creatinine less than 1.5 mg/dl or creatinine clearance greater than 60 ml/hr; SGOT and SGPT less than 4 times the upper limit of normal.

Patients must have an ANC greater than 2000/mm(3) and platelets greater than 100,000/mm(3).

Patients must be at least 18 years of age.

Patients of all racial and gender groups will be included.

Patients must not have received any prior gemcitabine, radiotherapy, or Herceptin therapy for pancreatic cancer.

Patients cannot receive concurrent hormonal or immunotherapy treatment for pancreatic cancer.

Patients cannot receive any anti-tumor therapy within 30 days of protocol eligibility and must have recovered from any prior treatment related toxicity.

Patients must not have evidence of distant metastases (e.g., peritoneal, carcinomatosis, liver metastases).

No concurrent second malignancy other than non-melanoma skin cancer or cervical carcinoma in situ.

Must not have medical conditions that preclude undergoing surgery or receiving therapy or follow up, or have psychiatric disease which would prevent adequate informed consent or render receiving this therapy unsafe.

No patients with an LV ejection fraction less than the lower limit of normal as determined at the Clinical Center, NIH.

Women must not be pregnant or nursing due to the unknown effects of this therapy on the unborn or nursing child.

Must not have received prior abdominal or pelvic radiation.

Must not have recent myocardial infarction (less than 6 months prior), unstable angina, or congestive heart failure (NYHA class III or IV).

Must not have active diseases which make the patient more susceptible to infection, including but not limited to AIDS, hepatitis, history of autoimmune disorders, because the experimental treatment being evaluated in this protocol may be unsafe in the absence of an intact immune system.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2000-06; Study Completion 2000-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Jessup JM, Steele G Jr, Mayer RJ, Posner M, Busse P, Cady B, Stone M, Jenkins R, Osteen R. Neoadjuvant therapy for unresectable pancreatic adenocarcinoma. Arch Surg. 1993 May;128(5):559-64. doi: 10.1001/archsurg.1993.01420170093014. PMID 8098206
- [Background] Weese JL, Nussbaum ML, Paul AR, Engstrom PF, Solin LJ, Kowalyshyn MJ, Hoffman JP. Increased resectability of locally advanced pancreatic and periampullary carcinoma with neoadjuvant chemoradiotherapy. Int J Pancreatol. 1990 Aug-Nov;7(1-3):177-85. doi: 10.1007/BF02924235. PMID 2081923
- [Background] Moertel CG, Frytak S, Hahn RG, O'Connell MJ, Reitemeier RJ, Rubin J, Schutt AJ, Weiland LH, Childs DS, Holbrook MA, Lavin PT, Livstone E, Spiro H, Knowlton A, Kalser M, Barkin J, Lessner H, Mann-Kaplan R, Ramming K, Douglas HO Jr, Thomas P, Nave H, Bateman J, Lokich J, Brooks J, Chaffey J, Corson JM, Zamcheck N, Novak JW. Therapy of locally unresectable pancreatic carcinoma: a randomized comparison of high dose (6000 rads) radiation alone, moderate dose radiation (4000 rads + 5-fluorouracil), and high dose radiation + 5-fluorouracil: The Gastrointestinal Tumor Study Group. Cancer. 1981 Oct 15;48(8):1705-10. doi: 10.1002/1097-0142(19811015)48:83.0.co;2-4. PMID 7284971